CLINICAL TRIAL: NCT05561933
Title: COVID-19 and the Healthy Minds Program for Educators II
Brief Title: Scaling Well-Being for Educators During COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Chan Zuckerberg Initiative (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2022-0313; IRB Approval Date: 08/16/2022 (Other: UW Madison); A483000 (Other: UW Madison)
Record Dates: First submitted 2022-09-27; First posted 2022-09-30 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-05

CONDITIONS: Anxiety; Depression
Keywords: Well-being
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Intervention Model Description: Random parallel assignment
Who Masked: Investigator, Outcomes Assessor
Masking Description: The investigator and data analyst will not know condition assignment until after data analyses are complete.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Choice Group (Placebo Comparator): Participants assigned to the Choice group will receive a list of digital (i.e., links to TED talks) and hard-copy (i.e., books) resources that focus on the science of well-being and may support well-being. It is up to participants whether and to what extent they choose to engage with these resources. A study library with 10 copies of each recommended book will be accessible to participants should they wish to read any of the suggested books. After follow-up testing, Choice group participants will be provided free access to the HMP training.
  Interventions: Behavioral: Healthy Minds Program Foundations Training
- Healthy Minds Program (HMP) Group (Experimental): Participants in the experimental arm will be assigned to the Healthy Minds Program Foundations training (HMP) which consists of 30-days of didactic and experiential content in a scientifically-derived model of well-being.
  A second random assignment will occur among intervention participants in which participants will receive the standard Foundations training or the Foundations training plus once per day push notifications (i.e., a micro-interventions) that provide a very brief opportunity to practice with the HMP content of that day. HMP participants will not be made aware of this second assignment.
  Interventions: Behavioral: Healthy Minds Program Foundations Training

INTERVENTIONS:
Behavioral: Healthy Minds Program Foundations Training — The HMP was developed by Healthy Minds Innovations at the UW Center for Healthy Minds, and is based on decades of research on well-being. The program is delivered through a smartphone application and consists of didactic ("learns") and experiential ("practice") components. Practice components involve contemplative practices such as mindfulness, loving-kindness, and gratitude practices. Each practice allows participants to choose duration (between 5-30 minutes). In addition to sitting style practices common in other meditation apps/programs, the HMP also provides instruction in active practices. Active practices engage the same skills as sitting practice, but focus on strengthening skills during daily routines. Learn components provide psycho-educational content about the science of well-being. HMP learns and practices are based on a four pillar model of well-being skills consisting of Awareness, Connection, Insight, and Purpose.

SUMMARY:
This study is a randomized controlled trial (RCT) of the four-week Healthy Minds Program (HMP) app Foundations training in employees of Jefferson County Public Schools (JCPS) in Louisville, KY. The study will enroll 1300 JCPS employees.

After completing the baseline assessment, participants will be randomly assigned to the intervention (i.e., the Healthy Minds Program App) or to a "Choice" control condition. HMP assigned participants will receive instructions and support in downloading and activating the app. Choice assigned participants will receive a list of resources that are focused on the science of well-being and happiness consisting of TED talk videos and books. 10 copies of each suggested book will be available for participants to check out. TED talk video links will be provided and are free to watch. Each week during the 4-week intervention period, participants in both conditions will complete the same weekly set of measures. Within two-weeks following the end of the intervention period, all participants will complete the post-test assessment. Approximately five to six months following post-test, participants will complete the follow-up assessment. In addition to study team collected data, the research team will receive from the district multiple years of student records (e.g., standardized assessments, attendance, disciplinary referrals) linked to teachers (teachers only, not other categories of employees who choose to participate).

The researchers predict that participants assigned to the intervention will demonstrate significantly reduced anxiety and depressive symptoms and significantly improved well-being after the intervention, and these improvements will persist at the follow-up (primary outcomes). It is hypothesized that baseline participant characteristics and early experience of the intervention will predict treatment adherence, study drop-out and outcomes, and that treatment engagement will moderate outcomes. In addition, the investigators predict that intervention period improvements on well-being skills assessed weekly will mediate long-term improvements on primary outcomes.

DETAILED DESCRIPTION:
This study is a conceptual replication of COVID and the Healthy Minds for Educators (NCT04426318). It will test whether training in well-being practices, using the Healthy Minds Program (HMP) app, is beneficial for employees in Jefferson County Public Schools (JCPS) in Louisville, Kentucky. The goal is to extend the prior study by recruiting a larger and more diverse sample of participants and examining whether intervening at the staff level positively affects student outcomes.

The HMP app approaches cultivating well-being by training psychological skills with clear mechanistic hypotheses. There is no single definition of well-being, but consensus exists that positive functioning beyond the absence of detrimental mental health symptoms is central. Building on related "eudaimonic" frameworks of psychological flourishing that identify qualities like environmental mastery, positive relations with others, and personal growth, this program targets brain-based skills that underlie the active cultivation of such qualities (e.g., regulating attention, empathic care, mental flexibility), and thus offers straightforward hypotheses about mechanisms of change. The cultivation of such skills aligns with the World Health Organization's definition of mental health, as a state of well-being in which an individual can work productively, cope with the normal stresses of life, contribute to his or her community, and realize his or her own abilities. Viewing well-being as dynamic and skill-based, as opposed to static and set, brings new optimism to cultivating well-being across the lifespan.

The HMP app involves mental exercises that are integrated into daily life, with an approach that parallels the way physical exercise becomes a part of healthy living. A minority of the population is both free of mental illness and high in well-being. This group flourishes mentally and physically (e.g., fewest days of missed work, healthiest psychosocial functioning, lowest risk of cardiovascular disease, lowest health care utilization). Troubling mental health trends in the opposite direction, however, underscore the need for training that bolsters and sustains well-being. National survey data recently revealed that 75% of Americans are significantly impacted by stress (e.g., anxiety, sleeplessness, fatigue), a new high since the survey's inception in 2007. Social divisiveness is an alarming new theme in these reports (59% identified this as a cause of stress), especially given rising trends of social isolation in which people report far fewer trusted confidants (this isolation is even more pronounced now with "safer at home" orders). Whereas mental health interventions have traditionally focused on treating serious mental disorders, this program advocates training and practicing skills even when an individual is relatively healthy. In this framework, exercising these skill sets bolsters well-being and fosters future resilience during inevitable periods of stress and loss. This program offers an innovative public health approach to caring for the mind. By investigating the underlying mechanisms, the investigators will understand whether this potentially transformative approach is viable.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18 years old and up
* Employee of participating district/state
* Smartphone or device that can download apps from Google Play or the iTunes app store

Exclusion Criteria:

* Individuals under 18 years old
* Significant meditation experience:

  1. Meditation retreat experience (meditation retreat or yoga/body practice retreat with significant meditation component)
  2. Regular meditation practice weekly for over 1 year OR daily practice within the previous 6 months
  3. Previous use of the HMP app.
* PROMIS depression score greater than 70

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 829 (Actual)
Dates: Start 2022-10-21 (Actual); Primary Completion 2023-07-30 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Change From Baseline on Psychological distress: Z-scored aggregate of Patient-Reported Outcomes Measurement Information System (PROMIS) Depression (a) and Anxiety (b) Scales, and the NIH Toolbox Perceived Stress v2.0 (c). | baseline, after weeks 1, 2, and 3 of the intervention, 4 weeks (post intervention), 20 weeks (5 months post-intervention)
  A and B: Adaptive 4-8 item self-report scale. C: 10-item self-report. Higher scores indicate greater symptoms of psychological distress.

SECONDARY OUTCOMES:
Well-being (WHO-5) | baseline, after weeks 1, 2, and 3 of the intervention, 4 weeks (post intervention), 20 weeks (5 months post-intervention)
  The World Health Organization Five Well-Being Index (WHO-5) is a short self-reported measure of current mental well-being (time frame the previous two weeks). The scale score range is 0 (lowest possible well-being) to 25 (highest possible well-being.
Change From Baseline on the Five Facet Mindfulness Questionnaire Act With Awareness and Non-react to Inner Experience Subscales | baseline, after weeks 1, 2, and 3 of the intervention, 4 weeks (post intervention), 20 weeks (5 months post-intervention)
  A measure of acting with mindful awareness and not reacting to experience. Total possible scores range from 8-40, with higher scores indicating greater levels of the facet of mindfulness. These constructs are specified as a mechanism of change.
Change From Baseline on the NIH Toolbox Loneliness Scale. | baseline, after weeks 1, 2, and 3 of the intervention, 4 weeks (post intervention), 20 weeks (5 months post-intervention)
  A measure of loneliness (i.e, lack of social connectedness). The total possible range in scores is 1-5, representing the average across all items; higher scores indicate greater levels of loneliness. This construct is specified as a mechanism of change.
Change From Baseline on the Lee Coronavirus Anxiety Scale (CAS) | baseline, 4 weeks (post intervention), 20 weeks (5 months post-intervention)
  The Coronavirus Anxiety Scale (CAS) is a brief mental health screener to identify probable cases of dysfunctional anxiety associated with the COVID-19 crisis. The scale score range is 0 (lowest possible anxiety) to 20 (highest possible anxiety).
Change From Baseline on the Perseverative Thought Questionnaire | baseline, 4 weeks (post intervention)
  Negative ruminative thinking will be measured with the Perseverative Thought Questionnaire. The total possible range in scores is 0-60, with higher scores indicating greater levels negative ruminative thinking.
Change From Baseline on the Growth Mindset Scale for Well-Being | baseline, after weeks 2, 4 weeks (post intervention), 20 weeks (5 months post-intervention)
  A measure of fixed versus incremental mindset regarding well-being. The average across items for a possible range in scores from 1-6 will be measured, with higher scores indicating greater levels of incremental views on well-being (i.e., it can be learned). This construct is specified as a mechanism of change.
Change from Baseline in Healthy Minds Index | baseline, after week 2, 4 weeks (post intervention)
  The HM Index is a 17-item questionnaire assessing qualities trained in the HMP app (awareness, connection, insight, purpose). It is scored on a 0- to 4-point Likert scale where 0 = a low amount (e.g., never, not at all, none of the time) and 4 = a higher amount (e.g., always, to the highest degree, all of the time) of a particular quality. Total scores for the four subscales range as follows: Awareness (0 to 16), Connection (0 to 24), Insight (0 to 12), Purpose (0 to 16) where higher scores indicate more of each quality.
Change from Baseline in Perceived Stress Scale | baseline, after weeks 1, 2, and 3 of the intervention, 4 weeks (post intervention), 20 weeks (5 months post-intervention)
  The Perceived Stress Scale is a 10-item scale where participants report their level of perceived stress (e.g., "In the last month, how often have you felt nervous and 'stressed'?"). It is scored on a 5-point Likert scale where 0 = "never" to 4 = "very often." Total scores range from 0 to 40 where higher scores indicate greater perceived stress.
Change from Baseline in Teacher Job Satisfaction Scale (TJSS-9) Questionnaire | baseline, after week 2, 4 weeks (post intervention), 20 weeks (5 months post-intervention)
  The Teacher Job Satisfaction Scale (Pepe, 2011) is a questionnaire aimed at measuring job satisfaction in educational contexts. The TJSS-9 is composed of three dimensions: satisfaction with co-workers (3 items), satisfaction with parents (3 items) and satisfaction with students' behaviors (3 items). Items are rated on a 5-point scale (1 = I am highly dissatisfied with this aspect of the school, 5 = I am highly satisfied with this aspect of the school).
Change in Baseline in Positive Administrative Support Questionnaire (Appreciation and Trust Attributes) | baseline, 4 weeks (post intervention), 20 weeks (5 months post-intervention)
  The Positive Administrative Support survey examines the effects of perceived administrative support on teacher stress, job satisfaction, and school commitment with intent to stay in the field. The appreciation subscale consists of 3 items with scale scores ranging from 0 (lowest appreciation) to 15 (highest appreciation). The trust subscale consists of 4 items with scale scores ranging from 0 (lowest trust) to 20 (highest trust).
Change in Baseline in Rumination About Work at Home Survey | baseline, after weeks 1 and 2, 4 weeks (post intervention), 20 weeks (5 months post-intervention)
  Participants express their perceptions of their work-home conflict with three statements scored on a five-point scale (1 = not at all true of me, 5 = very true of me). Higher scores indicate more work-home conflict.
Change in Baseline in Maslach Burnout Inventory (Emotional Exhaustion and Depersonalization Subscores) | baseline, week 4 (post intervention), 20 weeks (5 months post-intervention)
  Burn-out is a syndrome conceptualized as resulting from chronic workplace stress that has not been successfully managed. Participants will use a 7-point frequency scale (ranging from 0-never to 6-daily) to indicate the extent to which they experienced each item (e.g., "I feel emotionally drained from my work."). Higher scores indicate higher degrees of burnout.
Change in Baseline in Personal Wellbeing Index (PWI) | baseline, week 4 (post intervention), 20 weeks (5 months post-intervention)
  The PWI is a single question asking how satisfied the respondent feels in their life and personal circumstances on a Likert scale of 0 (no satisfaction at all) to 10 (completely satisfied), with higher scores indicating more satisfaction.
Change in Baseline in Sleep Quality | baseline, after weeks 1 and 2, 4 weeks (post intervention), 20 weeks (5 months post-intervention)
  Four items from the Pittsburgh Sleep Quality Index will be used to evaluate overall sleep quality, average nightly hours slept, use of sleep medications, and problems staying awake. All items except average nightly sleep are rated on a 1 (best) to 4 (worst) scale. The average nightly hours of sleep is scored so that >7 hrs a night (1), 6-7 hrs a night (2), 5-6 hrs a night (3), and <5 hrs a night (4). The four items are then averaged for an overall index of sleep quality.
Persistence in the profession | 12-18 months after baseline
  Using employment records provided by the district, investigators will compare the odds of continuing in the profession between the intervention and control groups in the 2023-2024 school year.
Change from baseline on reflection rings / circles | baseline, 4 weeks (post intervention), 20 weeks (5 months post-intervention)
  A gamified measure of allocentric circles measuring sense of connection. The task ask participants to move the degree to which two circles (one represents self, one an object) overlap as an indication of their feeling of connection with the object. Objects are others (e.g., friends, loved ones, parents, stranger) and things from the natural world (e.g., animals, eagle, trees). Rankings range from 0 (no overlap/no connection) t0 9 (complete overlap, indistinguishable). There is a total score (average of all items) as well as average scores on "others" and "natural world" items.
Change from baseline on experience sampling measure of satisfaction and mood at work and at home | baseline, 4 weeks (post intervention), 20 weeks (5 months post-intervention)
  A measure of satisfaction and mood at work and at home assessed 3 times a day, for 3 days. Scores on work life, job and home life satisfaction range from 1 (Not at all) to 5 (extremely) and scores on mood at work and mood at home range from 1 (very disatisfied) to 5 (very satisfied). Mood at work and home items rate the percentage of time a participants is in an irritable or bad mood at each place from 1 (0-25% of the time) to 4 (75-100% of the time).

OTHER OUTCOMES:
Digital Working Alliance Inventory | after weeks 1, 2, and 3 (intervention group only)
  A measure of working alliance in a digital environment that will be averaged across all items for a score range from 1 to 7, with higher scores reflecting higher levels of alliance. This construct will be used within the treatment arm as a predictor of engagement and outcomes.
Social Desirability (SDRS-5) | baseline
  SDRS measures an individual's tendency to portray a positive self-image when reporting pro-social behaviors. There are five items scored on a Likert scale from 1 (definitely true) to 5 (definitely false), with higher scores indicating a more positive self-image when reporting pro-social behaviors. This measure may be used a covariate.
Predictor of Drop-out Questionnaire | baseline
  The Predictor of Drop-out is a single question asking the respondent how likely they are to complete the study on a Likert scale of 1 (very unlikely) to 7 (very likely), with higher scores indicating lower prediction of drop-out. This construct will be used as a predictor of study completion.
Determinants of Meditation Practice Inventory-Revised (DMPI-R) | baseline
  The DMPI-R assesses perceived barriers to meditation among individuals without prior meditation experience. Items are scored on 5-point Likert-type scales (1 = strongly disagree, 5 = strongly agree). The scoring instructions are to sum all items to yield a total score (range = 12-60), with higher scores reflecting higher levels of perceived barriers to meditation. This construct will be used within the treatment arm as a predictor of engagement and outcomes.
Adverse Meditation Experiences Questionnaire | 4 weeks (post intervention), 20 weeks (5 months post-intervention)
  The Adverse Meditation Experiences questionnaire evaluates a participant's potentially negative experiences as a result of practicing meditation during the study. We will use 16-items from this scale to assess the propensity of participants who practiced meditation to experience challenge or distress, the intensity of the challenge/distress, the duration of the challenge/distress, and the degree to which these experience impacted functioning. Participants will rate their degree of confidence that meditation was the cause of their difficult experience as well as the degree to which they were glad to have practiced meditation in light of their answers to the prior questions.
Teacher effects on student change on standardized test scores | 6-months prior to baseline, baseline, 6-months, 18-months
  2022-2023 year students of participating teachers 2021-2022, 2022-2023, and 2023-2024 year standardized assessment scores
Teacher effects on student change on attendance | 6-months prior to baseline, baseline, 6-months, 18-months
  2022-2023 year students of participating teachers 2021-2022, 2022-2023, and 2023-2024 year attendance
Teacher effects on student change on disciplinary referrals | 6-months prior to baseline, baseline, 6-months, 18-months
  2022-2023 year students of participating teachers 2021-2022, 2022-2023, and 2023-2024 year disciplinary referrals

CONTACTS AND LOCATIONS:
Overall Officials: Matthew J Hirshberg, Principal Investigator — UW-Madison
Locations (1):
- Jefferson County Public Schools, Louisville, Kentucky, United States

IPD SHARING:
Plan to Share IPD: Yes
Prespecified hypotheses and analyses plans will be preregistered on osf.io prior to recruitment. De-identified study data will be posted on osf.io after publication of trial analyses. Code used in all publications will be available by request.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Study hypotheses and statistical analysis plans will be preregistered prior to enrollment and made publicly available at the time of relevant manuscript submissions. Analytic code will be made available following manuscript publication. De-identified study data will be made publicly available following manuscript publication. All public information will be accessible for an indefinite period of time.
Access Criteria: No access criteria

REFERENCES:
- [Background] Pilkonis PA, Choi SW, Reise SP, Stover AM, Riley WT, Cella D; PROMIS Cooperative Group. Item banks for measuring emotional distress from the Patient-Reported Outcomes Measurement Information System (PROMIS(R)): depression, anxiety, and anger. Assessment. 2011 Sep;18(3):263-83. doi: 10.1177/1073191111411667. Epub 2011 Jun 21. PMID 21697139
- [Background] Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. J Health Soc Behav. 1983 Dec;24(4):385-96. No abstract available. PMID 6668417
- [Background] Bech, P. (2004). Measuring the dimension of psychological general well-being by the WHO-5. Quality of Life Newsletter, 15-16.
- [Background] Maslach, C., Jackson, S. E., & Leiter, M. P. (1996). Maslach burnout inventory manual. Mountain View, CA: CPP. Inc., and Davies-Black.
- [Background] Crain TL, Schonert-Reichl KA, Roeser RW. Cultivating teacher mindfulness: Effects of a randomized controlled trial on work, home, and sleep outcomes. J Occup Health Psychol. 2017 Apr;22(2):138-152. doi: 10.1037/ocp0000043. Epub 2016 May 16. PMID 27182765
- [Background] Yu L, Buysse DJ, Germain A, Moul DE, Stover A, Dodds NE, Johnston KL, Pilkonis PA. Development of short forms from the PROMIS sleep disturbance and Sleep-Related Impairment item banks. Behav Sleep Med. 2011 Dec 28;10(1):6-24. doi: 10.1080/15402002.2012.636266. PMID 22250775
- [Background] Pepe A, Addimando L, Veronese G. Measuring Teacher Job Satisfaction: Assessing Invariance in the Teacher Job Satisfaction Scale (TJSS) Across Six Countries. Eur J Psychol. 2017 Aug 31;13(3):396-416. doi: 10.5964/ejop.v13i3.1389. eCollection 2017 Aug. PMID 28904592
- [Background] Lee SA. Coronavirus Anxiety Scale: A brief mental health screener for COVID-19 related anxiety. Death Stud. 2020;44(7):393-401. doi: 10.1080/07481187.2020.1748481. Epub 2020 Apr 16. PMID 32299304
- [Background] Britton WB, Lindahl JR, Cooper DJ, Canby NK, Palitsky R. Defining and measuring meditation-related adverse effects in mindfulness-based programs. Clin Psychol Sci. 2021 May 18;9(6):1185-1204. doi: 10.1177/2167702621996340. Epub 2021 Nov 1. PMID 35174010
- [Background] Brose, A., Raedt, R. D., & Vanderhasselt, M.-A. (2020). Eight items of the ruminative response scale are sufficient to measure weekly within-person variation in rumination. Current Psychology. https://doi.org/10.1007/s12144-020-00913-y
- [Background] Goldberg SB, Baldwin SA, Riordan KM, Torous J, Dahl CJ, Davidson RJ, Hirshberg MJ. Alliance With an Unguided Smartphone App: Validation of the Digital Working Alliance Inventory. Assessment. 2022 Sep;29(6):1331-1345. doi: 10.1177/10731911211015310. Epub 2021 May 18. PMID 34000843
- [Background] Baer RA, Smith GT, Lykins E, Button D, Krietemeyer J, Sauer S, Walsh E, Duggan D, Williams JM. Construct validity of the five facet mindfulness questionnaire in meditating and nonmeditating samples. Assessment. 2008 Sep;15(3):329-42. doi: 10.1177/1073191107313003. Epub 2008 Feb 29. PMID 18310597
- [Background] Cyranowski JM, Zill N, Bode R, Butt Z, Kelly MA, Pilkonis PA, Salsman JM, Cella D. Assessing social support, companionship, and distress: National Institute of Health (NIH) Toolbox Adult Social Relationship Scales. Health Psychol. 2013 Mar;32(3):293-301. doi: 10.1037/a0028586. PMID 23437856
- [Background] Devilly GJ, Borkovec TD. Psychometric properties of the credibility/expectancy questionnaire. J Behav Ther Exp Psychiatry. 2000 Jun;31(2):73-86. doi: 10.1016/s0005-7916(00)00012-4. PMID 11132119
- [Background] Hays, R. D., Hayashi, T., & Stewart, A. L. (1989). A five-item measure of socially desirable response set. Educational and Psychological Measurement, 49(3), 629-636.
- [Background] International Wellbeing Group (2013). Personal Wellbeing Index: 5th Edition. Melbourne: Australian Centre on Quality of Life, Deakin University
- [Background] Goldberg SB, Imhoff-Smith T, Bolt DM, Wilson-Mendenhall CD, Dahl CJ, Davidson RJ, Rosenkranz MA. Testing the Efficacy of a Multicomponent, Self-Guided, Smartphone-Based Meditation App: Three-Armed Randomized Controlled Trial. JMIR Ment Health. 2020 Nov 27;7(11):e23825. doi: 10.2196/23825. PMID 33245288
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771